CLINICAL TRIAL: NCT06491368
Title: Optimal Interval Between Consecutive Cesarean Sections: A Comparative Study on Maternal and Neonatal Outcomes
Brief Title: Optimal Interval Between Consecutive Cesarean Sections
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy, Lecturer of Obstetrics and Gynecology, Al-Azhar University
Other Study IDs: Obstet30624
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Section Complications
Keywords: Elective cesarean section; Time interval between consecutive cesarean sections
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Less than 18 months: This group consists of women who have had their previous cesarean section less than 12 months before the current scheduled elective cesarean section.
  Interventions: Procedure: Cesarean Delivery
- 18-24 months: This group includes women whose previous cesarean section was 12 to 24 months before their current scheduled elective cesarean section.
  Interventions: Procedure: Cesarean Delivery
- 25-36 months: This group is comprised of women who had their last cesarean section between 25 and 36 months prior to the current scheduled elective cesarean section.
  Interventions: Procedure: Cesarean Delivery
- 37-48 months: This group consists of women whose previous cesarean section occurred 37 to 48 months before the current scheduled elective cesarean section.
  Interventions: Procedure: Cesarean Delivery
- More than 48 months: This group includes women who had their last cesarean section more than 48 months before their current scheduled elective cesarean section.
  Interventions: Procedure: Cesarean Delivery

INTERVENTIONS:
Procedure: Cesarean Delivery — A Pfannenstiel abdominal incision is made. The skin and rectus sheath are transversely opened using sharp dissection, and the rectus sheath is separated from the underlying rectus abdominis muscles. The peritoneum is then longitudinally opened using sharp dissection. A transverse incision is made in the lower segment of the uterus, which is subsequently closed with two layers of continuous sutures. Both peritoneal layers are closed with continuous sutures. The fascia is closed using either continuous or interrupted sutures. Finally, the skin is closed with either interrupted sutures or a continuous intracutaneous suture.

SUMMARY:
The goal of this observational study is to determine the best time interval between consecutive cesarean sections and compare maternal and neonatal outcomes in women with a history of previous cesarean sections. The main questions it aims to answer are:

* What is the optimal time interval between consecutive cesarean sections for minimizing maternal intraoperative complications, blood transfusions, and intra- and postoperative bleeding?
* What are the differences in fetal and neonatal outcomes based on different time intervals between cesarean sections?

Participants will be divided into five subgroups based on the time interval since their last cesarean section: 0-12 months, 12-24 months, 25-36 months, 37-48 months, and more than 48 months. Each participant will undergo an elective cesarean section and provide data on maternal and neonatal outcomes.

Researchers will compare these subgroups to see if varying time intervals between consecutive cesarean sections affect maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-42 years.
* Full-term pregnant women more than 37 weeks gestation.
* Women with a history of at least one previous cesarean section, planning an elective repeated cesarean section.

Exclusion Criteria:

* Women with contraindications to cesarean section
* Those with emergency indications
* Multiple pregnancies
* Pre-existing maternal or fetal conditions affecting outcomes.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants who have undergone previous Cesarean section(s) and are scheduled for elective Cesarean section(s) as part of the study.
Study Population: The study population consists of 200 women who have undergone previous Cesarean sections and are scheduled for elective Cesarean sections. Participants are categorized into five groups based on the time interval since their last Cesarean section: Less than 18 months, 18-24 months, 25-36 months, 37-48 months, and more than 48 months. This study aims to compare maternal and neonatal outcomes across these different interval groups to determine the optimal interval between consecutive Cesarean sections for improving maternal and neonatal health outcomes.
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative complications | Withen the surgery.
  Occurrences of injuries to the bladder or bowel during surgery, injury of uterine artery, extension of uterine incision.

SECONDARY OUTCOMES:
Intraoperative and postoperative bleeding (quantify blood loss | withen the surgery and up to 24 hours after the sutgery.
  Measurement of blood loss before and after surgery using complete blood count (CBC).
Blood transfusions | withen the surgery and up to 24 hours after the sutgery.
  Instances of maternal blood transfusions during or after surgery.
ICU admissions | 1 week after the surgery.
  Number of mothers admitted to the Intensive Care Unit (ICU) postoperatively.
Fetal distress | during and 24 hours after the surgery.
  Instances of fetal distress noted during labor or delivery
Neonatal Apgar scores | 5 minutes after birth.
  Apgar scores measured at 1 minute and 5 minutes after birth, assessing newborn health.
NICU admissions | during and 24 hours after the surgery.
  Number of neonates admitted to the Neonatal Intensive Care Unit (NICU).
Neonatal morbidity and mortality | during and 2 weeks after the surgery.
  Incidence of health issues and deaths among newborns within a specific timeframe post-delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Hussein University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) from this study will be shared to facilitate transparency and further research. This includes anonymized data related to maternal and neonatal outcomes, as well as demographic and clinical variables collected during the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available after completion of the primary analysis and publication of the study results. Data sharing will commence within 6 months of publication and remain accessible for a minimum of 5 years to allow for secondary analyses and replication studies.
Access Criteria: Researchers interested in accessing IPD must submit a formal request detailing their research objectives, proposed analyses, and ethical approval from their institution's review board. Access will be granted based on the scientific merit of the proposed study and its alignment with the original research aims. Requests should be sent to the corresponding author.